CLINICAL TRIAL: NCT02359448
Title: Single-centre Open Label Exploratory Phase IIb Pilot Study of Exogenous Oral Melatonin for the Treatment of Nocturia in Adults With Parkinson's Disease
Brief Title: Melatonin for Nocturia in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0382
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease; Nocturia
MeSH Terms: conditions — Parkinson Disease; Nocturia | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melatonin (Experimental): Patients will be prescribed and dispensed from pharmacy sustained -release Melatonin (Circadin) 2mg. This will be taken every night for twelve weeks.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — An open label clinical trial of sustained-release Melatonin 2mg once daily for 6 weeks.
  Other Names: Circadin

SUMMARY:
This is an an open label clinical trial of sustained-release Melatonin 2mg once daily for 12 weeks in patients with Parkinsons's Disease reporting nocturia, defined as getting up regularly at night > twice to pass urine. The primary objective of this study is to evaluate the effects of exogenous melatonin on bother related to nocturia. Secondary objectives are to evaluate: 1) Mean night time urinary frequency 2)Volume of urine voided at night 3)Incontinence and other lower urinary tract symptoms (LUTS) 3)Quality of sleep 4) Quality of life 5) Sleep disturbance of partners 6)Safety

DETAILED DESCRIPTION:
This is a Phase IIb, open label single-site trial of sustained-release Melatonin 2mg in patients with PD, reporting nocturia, defined as getting up regularly at night > twice to pass urine. The primary objective of this study is to evaluate the effects of exogenous melatonin on bother related to nocturia. Secondary objectives are to evaluate: 1) Mean night time urinary frequency 2)Volume of urine voided at night 3)Incontinence and other lower urinary tract symptoms (LUTS) 3)Quality of sleep 4) Quality of life 5) Sleep disturbance of partners 6)Safety.

Patients will be asked to fill out questionnaires, diaries and to wear a wrist actiwatch for 2 weeks prior to starting melatonin and during the last 2 weeks of the 6 weeks treatment. A research nurse will telephone patients weekly whilst the patient is on Melatonin to enquire about medication use and any adverse events.

After taking consent, the investigator will take a history covering urinary symptoms, and causes for nocturia, e.g. medications. Participants will be examined and severity of PD assessed using Hoehn and Yahr staging and UPDRS (Unified Parkinson's Disease Rating Scale). Height, weight and supine/standing blood pressure will be recorded.

Urodynamics will be performed according to ICS Good Urodynamic Practice and will include uroflowmetry, bladder scan, filling cystometry and pressure flow study.

This pilot study aims to evaluate any effect that melatonin may have on nocturia related bother in Parkinson's Disease. Chi square test will be used to analyse change in bother related to nocturia (primary outcome) and number of nocturia episodes and questionnaire scores (Secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

1. Adults male and female(> 18 years) with clinically diagnosed PD according to the Brain Bank Criteria
2. Reporting nocturia to NMSQuest item 9 -"Getting up regularly at night to pass urine" and getting up to pass urine two or more times at night. Although the International Continence Society (ICS) defines nocturia as waking up at night one or more times to void, a recent population based study has shown that two voids or more is associated with bother and impaired health related quality of life.
3. Able to provide informed written consent

Exclusion Criteria:

1. Montreal Cognitive Assessment (MOCA) score < 26
2. History suggestive of REM sleep behaviour disorder
3. Congestive heart failure, liver failure or kidney failure as determined by medical history
4. Uncontrolled diabetes, or significant microalbuminuria in patients with diabetes
5. Using medications such as benzodiazepines and Z-drugs (e.g. Zaleplon, Zolpidem and Zopiclone)
6. Presence of urinary tract infection as determined by the clinician
7. Evidence for incomplete bladder emptying, i.e., post void residual urine of more than 100 mL as determined by ultrasound (bladder scan)
8. Presence of significantly enlarged prostate as determined by the clinician using the European Association of Urology (EAU) guidelines based on urodynamic findings
9. Females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
10. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment.
11. Females must not be breastfeeding.
12. Allergies to excipients of IMP
13. Smokers
14. Patient with autoimmune disease
15. Patients taking carbamazepine, rifampicin and cimetidine
16. Patients with rare hereditary problems of galactose intolerance, the LAP lactose deficiency or galactose malabsorption
17. Excessive alcohol consumption as defined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in bother related to nocturia as measured by a standardised validated questionnaire(ICIQ-N) | 6 weeks
  The primary outcome of this study is improvement on bother related to nocturia, as measured by the International Consultation on Incontinence Questionnaire Nocturia Module (ICIQ-N).

SECONDARY OUTCOMES:
Improvement in mean night time urinary frequency assessed from the frequency volume chart and a standardised validated questionnaire(ICIQ-N) | 6 weeks
Improvement in the Nocturnal polyuria index, percentage of volume of urine voided at night, calculated from the frequency volume chart. | 6 weeks
Improvement in overall lower urinary tract symptoms (LUTS), assessed by standardised validated questionnaires, ie. Urinary Symptom Profile | 6 weeks
Improvement on sleep disturbances, assessed using a standardised validated questionnaire, Pittsburgh Sleep Quality Index, sleep diary and Actigraphy | 6 weeks
Sleep disturbance in partners/careers assessed by sleep diary and Pittsburgh Sleep Quality Index | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jalesh Panicker, Principal Investigator — UCL
Locations (1):
- National Hospital for Neurology and Neurosurgery and UCL Institute of Neurology, London, United Kingdom